CLINICAL TRIAL: NCT06517537
Title: The Observational Study of Modified Aortic Root Enlargement Procedure in Aortic Stenosis Patients With Small Aortic Annulus
Brief Title: Modified Aortic Root Enlargement Procedure
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-2357
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-06

CONDITIONS: Small Aortic Annulus; Aortic Root Enlargement Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARE: The ARE group underwent modified ARE+AVR surgery
- TAVR: TAVR group undergoes routine TAVR surgery

SUMMARY:
This study is a prospective observational clinical trial, in which severe AS patients aged 50-70 years with SAA choose modified ARE or TAVR according to their wishes to investigate the safety and efficacy of modified ARE; Compare the incidence and clinical outcomes of moderate to severe PPM after modified ARE and TAVR surgery; Evaluate the feasibility of postoperative mid valve TAVR and explore the most ideal initial surgical plan for this type of patient from a full lifecycle perspective.

DETAILED DESCRIPTION:
Small aortic annulus (SAA), which is prevalently observed in patients with severe aortic stenosis (AS), constitutes a significant challenge in treatment and may give rise to post-operative prosthetic valve mismatch (PPM) and an elevated late mortality rate. The optimal approach for treating SAA remains controversial. Transcatheter aortic valve replacement (TAVR) has yielded superior valvular hemodynamic outcomes in patients with SAA; however, the incidence of PPM subsequent to surgery remains considerable. Aortic root enlargement (ARE) represents an effective solution for SAA, but the conventional method of aortic ring enlargement for ARE has restricted efficacy. In 2021, Yang Bo proposed an enhanced ARE approach, where the mitral curtain of the aortic valve was incised in an inverted Y-shape along the left non-coronary junction, enabling the enlargement of the number 3-5 of the aortic ring

ELIGIBILITY:
Inclusion Criteria:

* 1) Symptomatic severe AS patients aged 50-70 years who are planning to undergo biological valve replacement (diagnostic criteria for echocardiography are: mean transvalvular pressure gradient ≥ 40mmHg or flow velocity ≥ 4.0 m/s, aortic valve area (AVA) ≤ 0.8 cm2 or iEOA<0.5 cm2/m2) 2) Merge SAA (defined as mean aortic annulus diameter ≤ 23 mm measured by CT)

Exclusion Criteria:

* 1) High surgical risk, STS score>8% 2) Severe lesions in multiple coronary arteries requiring PCI or CABG 3) Simultaneous surgical intervention is required for severe mitral and tricuspid valve disease 4) Combining other complex cardiovascular diseases requires simultaneous surgical treatment 6) Combined severe pulmonary arterial hypertension or left ventricular dysfunction (LVEF<40%) 7) Severe respiratory, liver and kidney dysfunction, or other important organ dysfunction combined 8) Concurrent infective endocarditis in active phase 9) Previous history of cardiac surgery

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe AS patients aged 50-70 years with SAA can choose modified ARE or TAVR according to their wishes to study the safety and effectiveness of modified ARE; Compare the incidence and clinical outcomes of moderate to severe PPM after modified ARE and TAVR surgery; Evaluate the feasibility of postoperative mid valve TAVR and explore the most ideal initial surgical plan for this type of patient from a full lifecycle perspective.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of moderate PPM and severe PPM after surgery | Before discharge, 3 months after surgery, and 1 year after surgery
  Prospective collection of all echocardiographic data before surgery and upon discharge, measuring mean aortic valve area (EOA), mean transvalvular pressure gradient, and the degree and type of aortic regurgitation (AR). According to the patient's BSA calculation of iEOA, 0.65-0.85cm2/m2 is diagnosed as moderate PPM, and<0.65cm2/m2 is diagnosed as severe PPM.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China